CLINICAL TRIAL: NCT03882580
Title: Reporting, Evaluating, Preventing and Treating the Cardiotoxicity Induced by Anticancer Drugs During a Specific Cardio-oncology Consult and Follow up in Routine Care
Acronym: NEOCARDIO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Principal Investigator, Joe Elie Salem, Assistant director, clinical investigation center Paris Est, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: CIC1421-19-05
Record Dates: First submitted 2019-03-13; First posted 2019-03-20 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Cardiovascular Complication; Cardiovascular Insufficiency; Cardiac Complication; Oncologic Complications; Cardiac Insufficiency; Metabolic Disorder; Vascular Disorder; Cardiac Disorder
Keywords: anticancer drugs; cardiac toxicities; cardiovascular prevention; vascular toxicities; metabolic toxicities; adverse drug reactions
MeSH Terms: conditions — Heart Failure; Metabolic Diseases; Vascular Diseases; Heart Diseases; Cardiotoxicity; Drug-Related Side Effects and Adverse Reactions | interventions — Antineoplastic Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Anti-Cancer Agents — Drugs and treatments used in cancer inducing cardiovascular and metabolic side effects

SUMMARY:
Several Drugs used in routine care in oncology induce rare but often severe or fatal cardiovascular or metabolic side effects. This study will investigate, evaluate, report and treat the cardiovascular side effects of anticancer drugs, through a specific cardiovascular routine checkup and follow-up taking place in several Cardio-oncology programs throughout France. The different including centers will be: Assistance Publique - Hôpitaux de Paris (APHP.6: Pitié-Salpétrière, Saint Antoine and Tenon's hospitals, Paris, France).

DETAILED DESCRIPTION:
Several anticancer and supportive care drugs used in oncology have an impact on the cardiovascular and metabolic systems, leading to a wide range of cardiovascular and metabolic disorders and side effects. Those are poorly described, due to the evolution of the anticancer pharmacopeia, and recent recognition of these adverse events. This study will investigate the potential benefits of a specialized cardio-oncology check-up and follow-up in this context.

ELIGIBILITY:
Inclusion Criteria:

* Suffering a cancer
* Evaluated within a cardio-oncology program

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering (or having suffered) from a cancer
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients having a benefit after this specific cardio-oncology check up and follow up | 5 years

SECONDARY OUTCOMES:
Evaluating the overall survival of patients suffering from cardiovascular or metabolic side effect of oncology treatments | 5 years
All relevants staisticals associations between adverse events and anticancer drugs | 5 years
All relevant statistical associations between cardiovascular toxicities, and anticancer drugs | 5 years
All relevants statistical associations between cardiovascular side effects induced by oncology treatments , and other potentials kind of side effects induced by oncology treatments | 5 years
All relevant statistical associations between duration and type of treatement used to manage cardiovascular side effects induced by oncology treatments, and overall survival | 5 years
All relevants statistical associations between differential features of subgroups of patients, and the occurence of cardiovascular side effects induced by oncology treatments | 5 years
All relevant statistical associations between new therapies to treat or prevent the cardiovascular side effects induced by oncology treatments, and overall survival | 5 years
All relevant statistical associations between the pre therapeutic cardiovascular checkup and follow up for patients with cancer or history of cancer, and the occurence of cardiovascular toxicities of oncology treatments. | 5 years
All relevant statistical associations between metabolic toxicities, and anticancer drugs | 5 years
All relevants statistical associations between metabolic side effects induced by oncology treatments , and other potentials kind of side effects induced by oncology treatments | 5 years
All relevant statistical associations between duration and type of treatement used to manage metabolic side effects induced by oncology treatments, and overall survival | 5 years
All relevants statistical associations between differential features of subgroups of patients, and the occurence of metabloic side effects induced by oncology treatments | 5 years
All relevant statistical associations between new therapies to treat or prevent the metabolic side effects induced by oncology treatments, and overall survival | 5 years
All relevant statistical associations between the pre therapeutic metabolic checkup and follow up for patients with cancer or history of cancer, and the occurence of metabolic toxicities of oncology treatments. | 5 years

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - AP-HP, Saint-Antoine Hospital, Department of cardiology, Paris
  - AP-HP, Pitié-Salpêtrière Hospital, Department of Pharmacology, CIC-1421, Pharmacovigilance Unit, INSERM, Paris
  - AP-HP, Tenon Hospital, Department of Cardiology, Paris

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Salem JE, Allenbach Y, Vozy A, Brechot N, Johnson DB, Moslehi JJ, Kerneis M. Abatacept for Severe Immune Checkpoint Inhibitor-Associated Myocarditis. N Engl J Med. 2019 Jun 13;380(24):2377-2379. doi: 10.1056/NEJMc1901677. No abstract available. PMID 31189043
- [Derived] Dolladille C, Ederhy S, Allouche S, Dupas Q, Gervais R, Madelaine J, Sassier M, Plane AF, Comoz F, Cohen AA, Thuny FR, Cautela J, Alexandre J. Late cardiac adverse events in patients with cancer treated with immune checkpoint inhibitors. J Immunother Cancer. 2020 Jan;8(1):e000261. doi: 10.1136/jitc-2019-000261. PMID 31988143